CLINICAL TRIAL: NCT03550859
Title: Randomized, Open, Multicenter Study to Evaluate the Renal Function of HMG-CoA Reductase add-on in Chronic Kidney Disease Patients With Proteinuria
Brief Title: HMG-CoA Reductase add-on in Chronic Kidney Disease Patients With Proteinuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC030
Record Dates: First submitted 2018-05-09; First posted 2018-06-08 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Chronic Kidney Disease; Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Telmisartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duowell Tab. 40/10mg (Experimental): Telmisartan/Rosuvastatin 40/10mg qd for 48 weeks
  Interventions: Drug: Telmisartan/Rosuvastatin 40/10mg
- Micardis Tab. 40mg (Active Comparator): Telmisartan 40mg qd for 48 weeks
  Interventions: Drug: Telmisartan 40mg

INTERVENTIONS:
Drug: Telmisartan/Rosuvastatin 40/10mg — Telmisartan/Rosuvastatin 40/10mg qd for 48 weeks
  Arms: Duowell Tab. 40/10mg
Drug: Telmisartan 40mg — Telmisartan 40mg qd for 48 weeks
  Arms: Micardis Tab. 40mg

SUMMARY:
This study is to evaluate the renal function of HMG-CoA reductase add-on in chronic kidney disease patients with proteinuria.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 19 years
2. Chronic Kidney Disease (CKD) with CKD stage G2 or G3 and 300 mg/g ≤ urine PCR ≤ 3000 mg/g
3. Diagnosed with hypertension
4. Written informed consent
5. Patients who have not administered statin (including rosuvastatin) and hyperlipidemia treatment for at least 4 weeks prior to randomization

Exclusion Criteria:

1. Type I diabetes
2. Uncontrolled diabetic patients with HbA1c > 10% at screening
3. Hypertensive patients whose mean blood pressure was not controlled at 160/90 mmHg or more in triplicate despite the use of antihypertensive agents at the time of randomization
4. Calculated LDL-C ≥ 160 mg/dL at randomization
5. Patients who have taken RAS blockers (ACE inhibitor, ARB, and Aldosterone antagonist) for 4 weeks prior to randomization
6. Heart failure patients with NYHA class IV
7. Patients with acute and chronic liver disease, acute inflammation, hematologic abnormalities and cancer within the last 6 months
8. Patients with a history of cerebral blood cardiovascular complications (cerebral infarction, transient ischemic attack, myocardial infarction, unstable angina, coronary artery bypass, and percutaneous coronary intervention)
9. Patients taking immunosuppressive drugs
10. Patients undergoing eGFR <30 mL/min/1.73 m2 (CKD-EPI formula) or renal replacement therapy (dialysis or renal transplant) at screening
11. Patients with a change in eGFR (CKD-EPI formula) value showing a difference of more than 30% in the last 6 months at screening
12. Creatine kinase (CK) level ≥ 3x ULN (upper limit of normal range)
13. Patients who are pregnant or planning to become pregnant
14. Contraindications stated in the SPC of telmisartan or rosuvastatin
15. Those participating in other clinical trials for investigational products at screening
16. Patients deemed to be ineligible to participate in the trial by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of change from baseline to week 48 in Urine Protein to Creatinine Ratio (UPCR) | baseline, week 48

SECONDARY OUTCOMES:
Change from baseline to week 24 in UPCR | baseline, week 24
Change from baseline to week 24 and week 48 in Urine Albumin-to-Creatinine Ratio (UACR) | baseline, week 24, week 48
Change from baseline to week 24 and week 48 in estimated glomerular filtration rate (eGFR) | baseline, week 24, week 48
Change from baseline to week 48 in UPCR | baseline, week 48
Change from baseline to week 48 in high-sensitivity CRP (hs-CRP) | baseline, week 48
Change from baseline to week 48 in HOMA-insulin resistance (HOMA-IR) | baseline, week 48
Change from baseline to week 48 in 24hr urine protein | baseline, week 48
Proportion of subjects whose UPCR decreased by more than 30% at 48 weeks | baseline, week 48
Change from baseline to week 48 in MCP-1 (monocyte chemoattractant protein 1) | baseline, week 48
Change from baseline to week 48 in urinary 8-isoprostane | baseline, week 48
Change from baseline to week 48 in urine nephrin | baseline, week 48
Change from baseline to week 48 in type IV collagen | baseline, week 48
Proportion of subjects who received renal replacement therapy (dialysis or renal transplant) at 12, 24, 36, or 48 weeks | baseline, week 12, week 24, week 36, week 48

CONTACTS AND LOCATIONS:
Locations (16):
- South Korea (16):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Ansan Hospital, Ansan, Gyeonggido
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang
  - The Catholic University of Korea Incheon St.Mary's Hospital, Incheon
  - Presbyterian Medical Center, Jeonju
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - korea Universitiy Anam Hospital, Seoul
  - KyungHee Universitiy Hospital at Gandong, Seoul
  - SMG-SNU Boramae Medical Center, Seoul